CLINICAL TRIAL: NCT02241057
Title: A Randomized, Open-Label Study to Evaluate the Temperature Profile and Adhesion of an Air-Activated Adhesive-Backed Heat Patch in Healthy Volunteers
Brief Title: Investigational Air-Activated Adhesive-Backed Heat Patch (3-Cell)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chattem, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2014011
Record Dates: First submitted 2014-09-11; First posted 2014-09-16 (Estimated); Last update posted 2017-03-17 (Actual); Status verified 2016-01

CONDITIONS: Healthy
Keywords: temperature profile; air activated 3-cell patch; adhesion
MeSH Terms: conditions — Tissue Adhesions

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Temperature (Experimental): Evaluate the temperature profile of the air activated 3-cell patch during 8 hours of wear
  Interventions: Device: Investigational Air-Activated Adhesive-Backed Heat Patch (3-Cell); Other: Temperature Probe
- Adhesion (Experimental): Evaluate the adhesion with and without the presence of a temperature probe
  Interventions: Device: Investigational Air-Activated Adhesive-Backed Heat Patch (3-Cell)

INTERVENTIONS:
Device: Investigational Air-Activated Adhesive-Backed Heat Patch (3-Cell)
Other: Temperature Probe
  Arms: Temperature

SUMMARY:
This is an open-label study. A total of approximately 60 subjects will be randomly assigned to receive either the heat patch (30 subjects) with a temperature probe/skin reference probe or a heat patch (30 subjects) alone. The study will consist of 2 visits.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who complete an appropriately administered informed consent process that includes signing the consent form.
* Subjects 18-75 years old of either sex.
* Are of any skin type or race, providing the skin pigmentation will allow discernment of erythema;
* Subjects who are in good general health.
* Subjects who are willing and able to have the test products applied as directed, and comply with study instructions.
* Participants must be willing to restrict their activity for the 8 hour patch wear time.
* All participants agree to wear a t-shirt provided by the site for the entire 8 hour patch wear time.

Exclusion Criteria:

* Subjects who have a history of sensitivity to any of the test products or adhesion material.
* Subjects who are pregnant.
* Subject with excessive hair at the application sites, scar tissue, tattoo, or coloration that would interfere with placement of test product or skin assessment.
* Subjects with diabetes, rheumatoid arthritis, poor circulation or have any clinically significant chronic illness.
* Subjects with active dermatitis (including sunburn) in the treatment area, or other visible dermatological disease which, in the investigator's opinion, might interfere with the response to the test products or interfere with the skin assessments associated with the test products.
* Have history of significant dermatologic cancers (eg, melanoma, squamous cell carcinoma).
* Subjects who have used topical dermatological products in the application area within 24 hours prior to the test product application.
* Subject using a concomitant medication that, in the investigator's opinion, could interfere with the interpretation of study results. Examples of such drugs include non-steroidal anti-inflammatory drugs (NSAIDs, e.g., aspirin), topical or systemic corticosteroids, and cold/cough products containing antihistamines and/or either phentolamine, pseudoephedrine or phenylpropanolamine.
* Subjects who have received an investigational medication or device within 30 days prior to enrolment into this study.
* Subjects who are currently participating in an investigational study.
* Subject who are known to be noncompliant or are unlikely to comply with the requirements of the study protocol (e.g., due to alcoholism, drug dependency, mental incapacity) in the opinion of the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2014-09; Primary Completion 2014-09 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Patch Temperature | 8 hours
  The temperature of the patch will be monitored by the use of a probe placed under the patch and recorded for the duration of the study.
Patch Adhesion | 8 hours
  Patch adhesion will be recorded for the duration of the study.

CONTACTS AND LOCATIONS:
Overall Officials: Ellen Bonagua, MD, Principal Investigator — Chattem, Inc.
Locations (1):
- Wilkins Research, Chattanooga, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No